CLINICAL TRIAL: NCT05204290
Title: A Pilot Study of Combined Decompressive Spine Radiosurgery and Pembrolizumab in Patients With High-Grade Epidural Disease
Brief Title: Study of Combined Decompressive Spine Radiosurgery and Pembrolizumab
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Low accruals
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00078836; WFBCCC 03321 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-07

CONDITIONS: Epidural Spinal Tumors; Cancer
MeSH Terms: conditions — Epidural Neoplasms; Neoplasms | interventions — pembrolizumab; Radiosurgery; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stereotactic Body Radiotherapy and Pembrolizumab Treatment (Experimental): MRI scans of your spine (before treatment, 2 months after treatment, and 6 months after treatment) and immunotherapy with Pembrolizumab
  Interventions: Drug: Pembrolizumab; Radiation: Stereotactic Body Radiation Therapy; Other: Blood draws

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be delivered at the discretion of the patient's medical oncologist within 6 weeks after finishing SBRT. If a patient is already receiving pembrolizumab at the time of enrollment, then SBRT should not start sooner than 5 days after the last pembrolizumab infusion.
Radiation: Stereotactic Body Radiation Therapy — patients will undergo CT simulation and will be immobilized in either a BodyFix® or long thermoplastic mask depending on the location of the lesion. 1.25mm slices will be acquired. Dose and fractionation will be at the discretion of the treating radiation oncologist (as will the constraint to the spinal cord).
Other: Blood draws — Patients will have a blood draw at baseline and at 2-months post-SBRT, and 6 months post-stereotactic body radiation therapy.

SUMMARY:
The purpose of this research study is to find out what effects (good and bad) Pembrolizumab and radiosurgery have on participants with high-grade epidural disease of the spine.

DETAILED DESCRIPTION:
Primary Objective: To determine the feasibility of patients completing stereotactic body radiation therapy and at least one (1) cycle of Pembrolizumab.

Secondary Objectives:

* Evaluate the radiographic response after decompressive stereotactic body radiation therapy and Pembrolizumab by calculating the improvement in thecal sac patency (see 5.2.1).
* Evaluate accrual rate,
* Evaluate pain relief.
* Evaluate quality of life.
* Evaluate cumulative incidence of adverse events.
* Evaluate potential correlative blood biomarkers.

ELIGIBILITY:
Inclusion Criteria :

* Pathologic diagnosis of cancer, confirmed by review of pathology report.
* Epidural disease seen on MRI at 1 vertebral level or 2 contiguous vertebral level.
* Synchronous and metachronous sites of disease allowed.
* Patient with expected life span of ≥ 3 months.
* Deemed eligible for stereotactic body radiation therapy and pembrolizumab after multi-disciplinary review. The multi-disciplinary review will be conducted virtually via our Spinal Oncology Group (SPOG) Wake Forest e-mail listserv. Members of the distribution list include neurosurgeons, orthopedic surgeons, interventional radiologists, radiologists, and radiation oncologists. This group meets monthly via Webex and in the interim, cases are routinely reviewed using encrypted emails via the listserv. Because we will not be able to wait for a month meeting to enroll patients on study, we anticipate needing to review these patients via the listserv. The electronic review will serve as documentation of multi-disciplinary review.
* Patients currently being treated with pembrolizumab or anticipated to receive at least one dose of pembrolizumab within six weeks after finishing stereotactic body radiation therapy.
* Patients who have received prior immunotherapy are allowed.
* Age equal or greater than 18.
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria:

* Prior radiation therapy or surgery to index lesion.
* Patients with lymphoma, multiple myeloma, germinomas, seminomas, Wilm's tumors, and Ewing's sarcomas will be excluded.
* Muscle strength of ≤ 3 out of 5 on neurologic exam that correlates with level of the involved spinal cord.
* Retropulsed compression fracture.
* Patients with a contraindication to pembrolizumab.
* Patients may not be receiving any other investigational agents.
* Patients with symptomatic, brain metastases, as determined by the study PI, that could confound the neurologic exam, should be excluded.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because both radiation and pembrolizumab can be harmful to the developing fetus. Because there is an unknown but potential risk for adverse events, pregnant women are not allowed to participate in this study, in nursing infants secondary to treatment of the mother with pembrolizumab, breastfeeding should be discontinued.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants Completing Stereotactic Body Radiation Therapy and One Cycle of Pembrolizumab | 6 months
  A 95% confidence interval for the primary outcome, the feasibility of patients completing stereotactic body radiation therapy and at least one cycle of Pembrolizumab, will be calculated.

SECONDARY OUTCOMES:
Change Thecal Sac Patency - (Percentage) | at 2 months and 6 months after intervention
  The percentage of thecal sac patency, which will be calculated as the ratio of the thecal sac area at the level of greatest epidural disease to the estimated pre-compression thecal sac area. The estimated pre-compression thecal sac area will be calculated by averaging the area of the thecal sac at one spinal level above and one spinal level below the level of the compression.
Accrual Rate | Every 2 months, up to 20 months
  Number of enrolled per month on the study intervention.
Number of Participants Experiencing Improvement in Pain - Numeric Pain Rating Scale (NPRS) | At baseline and up to 20 months
  Using the Numeric Pain Rating Scale the number of participants that experience a clinically significant improvement in pain defined as either a 33% decrease in pain score or an absolute decrease from baseline of 2 points. Scores range from 0-10 points, with higher scores indicating greater pain intensity.
Quality of Life - European Organization for Research and Treatment of Cancer QoL Group Bone Metastases Module (QLQ-BM22) | Baseline, 2 months and 6 months
  The 22-item EORTC QLQ-BM22 questionnaire assesses disease symptoms related to bone metastasis, including painful sites, functional interference, painful characteristics, and psychosocial aspects as multi-item scales. Scaled items from one (not at all) to four (very much). Score range is from 0 to 100. A higher score in the case of symptom scales is indicative of greater distress, while a higher score in the case of functional scales indicates greater functional ability.
Incidences of Compression Fractures | 1 month after intervention and 6 months after intervention
  New or worsening after stereotactic body radiation therapy, rate of pain flare by physician assessment and cumulative incidences of radiation myelitis will be assessed. Radiation myelitis will be defined by the study PI using clinical and radiographic techniques will be calculated. For discrete variables, the proportions and counts will be calculated for each visit. For continuous variables, means, standard deviations, medians, the first quartiles, the third quartiles, and ranges will be calculated for each visit. The 95% confidence intervals will be also estimated
Changes in Plasma | At baseline, 2 months and 6 months after intervention
  Plasma will be tested for histamine, Calcitonin gene-related peptide (CGRP), and substance P which will characterize bone turnover markers, specifically for N-terminal propeptide of type 1 procollagen (P1NP; bone formation) and C-terminal telopeptide of type 1 collagen (CTX; bone resorption). For discrete variables, the proportions and counts will be calculated for each visit. For continuous variables, means, standard deviations, medians, the first quartiles, the third quartiles, and ranges will be calculated for each visit. The 95% confidence intervals will be also estimated

CONTACTS AND LOCATIONS:
Overall Officials: Christina K Cramer, MD, Principal Investigator — Wake Forest Baptist Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT05204290/ICF_000.pdf